CLINICAL TRIAL: NCT05988307
Title: Effect Of Percussion Massage Gun On Hamstrings Flexibility In Patients With Knee Osteoarthritis.
Brief Title: Effect of Percussion Massage Gun on Hamstrings Flexibility.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, heba mohamed moawed EL-berkawy, demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: percussion gun on Knee OA
Record Dates: First submitted 2023-07-30; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- receive percussion massage gun and conventional physical therapy program (Experimental)
  Interventions: Device: Percussion massage gun
- receive conventional physical therapy program only for knee osteoarthrities (Other)
  Interventions: Device: Percussion massage gun

INTERVENTIONS:
Device: Percussion massage gun — Percussion massage gun on hamstrings flexibility in patients with knee Osteoarthritis.
  Other Names: conventional physical therapy program

SUMMARY:
The purpose of this study would be to investigate:

* The effect of using percussion massage gun on Hamstring flexibility in patients with knee osteoarthritis.
* The effect of using percussion massage gun on pain in patients with knee osteoarthritis.
* The effect of using percussion massage gun on ROM in patients with knee osteoarthritis.
* The effect of using percussion massage gun on knee function in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is present in about 65% of people with knee pain aged 50 years or older. The condition is associated with knee pain and reduced function and those with progression of tibiofemoral OA. OA are at increased risk of both incidence and Approximately 11 percent of adults with knee osteoarthritis need help with personal care.

Conservative treatment consists of medication and various forms of physiotherapy including heat, massage, electrotherapy and exercises.. The hamstring muscle group have tendency to shorten and the tightening results in increased patello-femoral compressive force, which may eventually lead to patello-femoral syndrome often associated with osteoarthritis .

Percussion Therapy is a relatively new technique that uses a mechanical system, such as the massage gun, to provide percussion massage. The application of percussive massage gun activates the Golgi tendon organ, which triggers a relaxation response, improving circulation and nutrition to the tissue, and reducing tightness and improving flexibility, It also reduces pain perception through the pain gait theory process .

Currently there are no evidence based clinical guidelines for the use of mechanical percussion devices. Further laboratory-based and clinical outcomes studies are needed to best guide clinical practice regarding these devices; however, research should also be informed based on how the devices are utilized by clinicians when providing care to patients. Understanding the knowledge and current trends in the use of mechanical percussion devices among health care professionals may help guide researchers in developing guidelines for research and/or practice. Thus, the purpose of this study was to document the knowledge, clinical application methods, and use of mechanical percussion devices.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age - 40 years to 60 years patients of chronic knee OA (Culvenor et al., 2019).

  2. Patients with BMI < 30 kg/m² (not being classified as obese) 3. Patients who are able to walk with painful knee OA without assistive devices.

  4. Patients with knee pain intensity level at least >3 cm on a 10 cm VAS scale in activities such as going up-and downstairs, sitting and squatting.

Exclusion Criteria:

1. Radiated pain from low back pain.
2. Patients with no radiographic evidence of knee OA or with mild OA (grade I according to K/L classification) or with severe OA (grade IV according to K/L classification).
3. Loss of joint play in tibiofemoral and patellofemoral articulations.
4. Lower extremity fracture and surgery or trauma to the knee joint.
5. Neurological deficit or movement disorder related to lower limb.
6. Those who were athletes or who had been treated with physiotherapy or medications during the previous 6 weeks

   -

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
hamstring flexibility | baseline (1 month )
  measuring flexibility of hamstrings through sit and reach test and active knee extension

SECONDARY OUTCOMES:
measuring pain | baseline (1 month )
  through visual analogue scale .
measuring Function | baseline (1 month)
  through WOMAC questionnaire.

REFERENCES:
- [Background] Alghadir A, Anwer S, Iqbal ZA, Alsanawi HA. Cross-cultural adaptation, reliability and validity of the Arabic version of the reduced Western Ontario and McMaster Universities Osteoarthritis index in patients with knee osteoarthritis. Disabil Rehabil. 2016;38(7):689-94. doi: 10.3109/09638288.2015.1055380. Epub 2015 Jun 11. PMID 26066566
- [Background] 49. Lakhwani, M., & Phansopkar, P. (2021). Efficacy of Percussive Massage versus Calf Stretching on Pain, Range of Motion, Muscle Strength and Functional Outcomes in Patients with Plantar Fasciitis-A Research Protocol. Journal of Pharmaceutical Research International, 233(44B), 532-539.